CLINICAL TRIAL: NCT00322114
Title: Mechanism of Prostate Cancer Prevention by Lycopene
Brief Title: Lycopene in Preventing Prostate Cancer in Healthy Participants
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Illinois at Chicago (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Prevention
Other Study IDs: CDR0000468031; UIC-2004-0217
Record Dates: First submitted 2006-05-03; First posted 2006-05-04 (Estimated); Last update posted 2013-09-20 (Estimated); Status verified 2009-07

CONDITIONS: Prostate Cancer
Keywords: prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Lycopene

ARMS (3):
- Arm I (Experimental): Participants receive an oral tomato dietary supplement containing lycopene twice daily for 3 weeks.
  Interventions: Dietary Supplement: lycopene
- Arm II (Experimental): Participants receive an oral tomato dietary supplement containing lycopene at a higher dose twice daily for 3 weeks.
  Interventions: Dietary Supplement: lycopene
- Arm III (Placebo Comparator): Participants receive oral placebo twice daily for 3 weeks.
  Interventions: Other: placebo

INTERVENTIONS:
Dietary Supplement: lycopene — Given orally
  Arms: Arm I; Arm II
Other: placebo — Given orally
  Arms: Arm III

SUMMARY:
RATIONALE: Chemoprevention is the use of certain drugs or substances to keep cancer from forming, growing, or coming back. The use of lycopene, a substance found in tomatoes, may keep prostate cancer from forming.

PURPOSE: This randomized clinical trial is studying how well lycopene works in preventing prostate cancer in healthy participants.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine whether lycopene supplementation affects percent free and bound prostate-specific antigen (PSA) in healthy participants.

Secondary

* Determine whether lycopene reduces oxidative stress in these participants, as indicated by lipid peroxidation assay.
* Determine whether a 21-day washout period is sufficient to return lycopene, PSA, and lipid peroxidation products to baseline.

OUTLINE: This is a randomized, placebo-controlled study. Participants are randomized to 1 of 3 treatment arms.

* Arm I: Participants receive an oral tomato dietary supplement containing lycopene twice daily for 3 weeks.
* Arm II: Participants receive an oral tomato dietary supplement containing lycopene at a higher dose twice daily for 3 weeks.
* Arm III: Participants receive oral placebo twice daily for 3 weeks. Urine and blood samples are collected on days 0, 21, and 42.

PROJECTED ACCRUAL: A total of 150 participants will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Healthy participants
* No existing prostate disease

PATIENT CHARACTERISTICS:

* Able to supply blood and urine samples
* Able to answer demographic and dietary recall questionnaires
* No hospital inpatients
* Not allergic to tomatoes or tomato products
* Not abusing alcohol or non-prescribed drugs
* No existing gastrointestinal disease or cancer

PRIOR CONCURRENT THERAPY:

* At least 2 weeks since prior lycopene (in supplement form)
* No concurrent participation in another clinical trial

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2006-02; Primary Completion 2009-02 (Estimated)

PRIMARY OUTCOMES:
Measurement of changes in percent free and total serum prostate-specific antigen (PSA) induced by lycopene

CONTACTS AND LOCATIONS:
Overall Officials: Richard B. van Breemen, PhD, Principal Investigator — University of Illinois at Chicago
Locations (1):
- University of Illinois Cancer Center, Chicago, Illinois, United States